CLINICAL TRIAL: NCT02121691
Title: Appalachia Community Cancer Network II Centers for Reducing Cancer Disparities: Faith-Based Initiative to Promote Health in Appalachia
Brief Title: Faith-Based Initiative to Promote Health in Appalachia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Dignan, PhD (Other)
Responsible Party: Sponsor-Investigator, Mark Dignan, PhD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-085; NCI-2013-01400 (Other: NCI CTRP)
Record Dates: First submitted 2014-04-18; First posted 2014-04-23 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Cancer; Obesity
Keywords: Cancer; Obesity; Body Mass Index
MeSH Terms: conditions — Neoplasms; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Walk by Faith (Experimental): Intervention arm
  Interventions: Behavioral: Walk by Faith
- Comparison (No Intervention): Non-intervention arm

INTERVENTIONS:
Behavioral: Walk by Faith — The Walk by Faith program is aimed at increasing physical activity and improving healthy eating to reduce or maintain healthy BMI among members of the churches.
  Arms: Walk by Faith

SUMMARY:
The project will target two behavioral causes of obesity: a sedentary lifestyle and an unhealthy diet. The goal is to test a faith-based intervention among men and women who are members of participating Appalachian churches.

The primary hypothesis being tested in this project is: The change in body mass index from baseline to one year follow-up in intervention churches will be greater than among comparison churches, such that the differential change will be negative on average.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Member of the participating church who has attended services at least 4 times in the past 2 months
* resident of an Appalachia county
* Able bodied (no contraindications to physical activity and no dietary restrictions that are part of a medically prescribed diet for weight loss or formal weight loss program)
* Able to read and write in English
* Have a BMI indicating that they are overweight (BMI > or = 25.0, assessed during biometric measurement)
* Under 400 pounds (per self-report and confirmed during biometric measurement)
* Not planning to move out of the area within the next year
* Does not reside in nursing facility or residential home
* If female, is not pregnant, breastfeeding or less than 9 months post-partum and does not intend to become pregnant during the study
* Able to provide informed consent.

Exclusion Criteria:

* Does not meet Inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in body mass index from baseline to one year follow-up | Baseline, month 12

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dignan, PhD, MPH, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (5):
- United States (5):
  - Markey Cancer Center, Lexington, Kentucky
  - Ohio State University, Columbus, Ohio
  - Penn State University, University Park, Pennsylvania
  - Virginia Tech, Blacksburg, Virginia
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Derived] Zhang X, Shoben A, Felix AS, Focht BC, Baltic RD, Paskett ED. The mediating role of social support in behavioral changes and weight loss outcomes among overweight Appalachian adults. J Behav Med. 2025 Apr;48(2):360-372. doi: 10.1007/s10865-025-00555-0. Epub 2025 Feb 9. PMID 39924605